CLINICAL TRIAL: NCT06683937
Title: Evaluation of Direct Antiviral Treatments Against SARS-CoV-2 in Immunocompromised Patients With Covid-19. A G2i Study, National Multicenter Observational and Retrospective From June 2023 to April 2024
Acronym: COV-ID
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241194
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Immunocompromised Patients; SARS-CoV-2 Disease
Keywords: Immunocompromised patients; SARS-CoV-2 disease; Mono- or dual therapy with nirmatrelvir/ritonavir or remdesivir
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Adult patients at very high risk of severe SARS-CoV-2 disease, hospitalized for SARS-CoV-2 infection from June 2023 to April 2024.
  Interventions: Other: Collection of data from the patient's medical file

INTERVENTIONS:
Other: Collection of data from the patient's medical file — Collection of data from the patient's medical file

SUMMARY:
Due to the lower virulence of circulating Omicron variants and the high seroprevalence of anti-SARS-CoV-2 antibodies, the incidence of cases and deaths related to the SARS-CoV-2 virus has significantly decreased in recent months worldwide. However, these infections remain a major public health problem in severely immunocompromised patients, who have decreased vaccine efficacy and are at higher risk of persistent SARS-CoV-2 viral shedding, relapses, secondary invasive fungal infection, intensive care unit hospitalization, and death than non-immunocompromised patients.

The research concerns adult patients at very high risk of severe SARS-CoV-2 disease, suffering from SARS-CoV-2 having resulted in hospitalization in a center participating in the study in France between June 1, 2023 and April 1, 2024 and having received mono- or dual therapy with nirmatrelvir/ritonavir or remdesivir in order to carry out an evaluation of direct antiviral treatments against SARS-CoV-2 in these immunocompromised patients suffering from Covid-19.

The study consists of collecting patient care data from the medical record. Patients will be identified by practitioners at each participating French center.

DETAILED DESCRIPTION:
Due to the lower virulence of circulating Omicron variants and the high seroprevalence of anti-SARS-CoV-2 antibodies, the incidence of cases and deaths related to the SARS-CoV-2 virus has significantly decreased in recent months worldwide. However, these infections remain a major public health problem in severely immunocompromised patients, who have decreased vaccine efficacy and are at higher risk of persistent SARS-CoV-2 viral shedding, relapses, secondary invasive fungal infection, intensive care unit hospitalization, and death than non-immunocompromised patients.

The research concerns adult patients at very high risk of severe SARS-CoV-2 disease, suffering from SARS-CoV-2 having resulted in hospitalization in a center participating in the study in France between June 1, 2023 and April 1, 2024 and having received mono- or dual therapy with nirmatrelvir/ritonavir or remdesivir in order to carry out an evaluation of direct antiviral treatments against SARS-CoV-2 in these immunocompromised patients suffering from Covid-19.

Identifying an effective anti-SARS-CoV-2 therapeutic strategy is a real challenge in severely immunocompromised patients because clinicians are faced with chronic carriage and serious complications in these patients, as well as drug interactions with immunosuppressive treatments, the emergence of resistance and the absence of recommendations.

The data currently available in the literature remain heterogeneous and sometimes without sufficient level of evidence. However, some teams have reported in this population the efficacy of repeated or prolonged treatment with nirmatrelvir/ritonavir or even multitherapies combining several antiviral treatments and/or combinations of monoclonal antibodies on persistent carriage of the virus. Thus, some centers recommend prolonged antiviral treatments combining 5 to 10 days of remdesivir with 10 days of nirmatrelvir/ritonavir.

Nirmatrelvir/ritonavir and remdesivir are the currently available antiviral therapies that are still effective against circulating Omicron virus subvariants. It therefore seems important to have more data on their efficacy in monotherapy, dual therapy, or in the case of prolonged treatment.

The study consists of collecting patient care data from the medical record. Patients will be identified by practitioners at each participating French center.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with SARS-CoV-2 in France, treated in a center participating in the study
* Symptomatic patients for Covid-19 who have received mono- or dual therapy with nirmatrelvir/ritonavir or remdesivir
* SARS-CoV-2 positive by PCR on nasopharyngeal swab, ECBC or bronchoalveolar fluid
* Hospitalization in a ward or day hospital for SARS-CoV-2 infection
* Patients at very high risk of severe form of SARS-CoV-2

  * Aggressive lymphomas (all types)
  * Acute lymphocytic leukemia
  * Acute myeloid leukemia
  * Acute promyelocytic leukemia
  * T-cell prolymphocytic leukemia
  * Primary lymphoma of the central nervous system
  * Stem cell transplant
  * Light chain amyloidosis
  * Chronic lymphocytic leukemia
  * Multiple myeloma
  * Hematopoietic stem cell transplant
  * Solid organ transplant
  * Being on the waiting list for an organ transplant
  * Primary immunodeficiency;
  * HIV patients with CD4 <200/mm3 or with a detectable viral load
  * Lymphopenia <200/mm3
  * Neutropenia <1000/mm3 for > 1 week
  * Patients receiving long-term immunosuppressive treatment (period of at least 3 months during treatment during infection) with:
* anti-CD20 antibodies
* anti-JAK
* BTK inhibitors
* azathioprine
* cyclophosphamide
* methotrexate
* mycophenolate mofetil
* CAR-T cell gene therapy
* bi-phenotypic therapeutic antibodies
* tacrolimus
* sirolimus
* long-term corticosteroids (prednisone equivalent dose >5mg for 3 months)

Exclusion Criteria:

* Opposition formulated (following receipt of the study information note)
* Patients who received convalescent plasma as first-line treatment for SARS-CoV-2 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients at very high risk of severe SARS-CoV-2 disease, hospitalized for SARS-CoV-2 infection from June 2023 to April 2024 in France.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical evolution of immunocompromised patients receiving remdesivir and/or nirmatrelvir/ritonavir as curative treatment for COVID-19 | 37 days
  Evolution of the patient's modified (suitable for immunocompromised patients) Ordinal Scale for Clinical Improvement (OSCI) of the World Health Organization (WHO) (score from 0 - non infected patient to 8 - deceased patient) from the initiation of treatment to 30 days (+7 days) following the first line of therapy.

SECONDARY OUTCOMES:
Mortality at 30 days of diagnosis | 30 days
  Mortality at 30 days of diagnosis
Tolerance of antiviral treatments against SARS-CoV-2 | 6 months
  Rate of serious side effects within 6 months (grade 3 and 4 on adverse event scale).
Evaluate virological evolution | 60 days
  Decrease or negativity of PCR between D2 and D30 following the first line of anti-SARS-CoV-2 therapy, then at D60.
Evaluate radiological evolution | 90 days
  Reduction or disappearance of radiological lung lesions after the first line of therapy.
Clinical relapse at discharge from hospital, at D30 and D60 | 90 days
  Modified (suitable for immunocompromised patients ) OSCI score (Ordinal Scale for Clinical Improvement of the World Health Organization, score from 0 - non infected patient to 8 - deceased patient)at hospital discharge, D30 and D60. Maximum modified OSCI score between H48 and D30.
Identified factors associated with favorable evolution | 90 days
  Description of clinical evolution adjusted for age and other variables of interest.
Infectious complications and secondary non-infectious complications | 90 days
  Incidence of infectious complications (aspergillosis and bacterial infections) and secondary non-infectious complications.
  Collection of the following elements:
  * Use of a second line of therapy (antivirals and plasma therapy) specifying the time after the first line
  * occurrence of complications during the initial hospitalization after the first line of therapy: pulmonary embolism, hospitalization in the Intensive Care Unit, probable or proven invasive fungal infections (aspergillosis, mucormycosis with initiation of antifungal treatment), bacterial infection (antibiotics initiated)
  * persistence of viral carriage (> 3 weeks and >8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Cléa Melenotte, M.D., Principal Investigator — Assistance Publique - Hôpitaux de Paris; Clémentine de La Porte, M.D., Study Director — Assistance Publique - Hôpitaux de Paris
Locations (16):
- France (16):
  - CHU Angers, Angers
  - CHU Caen, Caen
  - Hôpital Pasteur, Colmar, Colmar
  - CHD Vendée (La Roche sur Yon), La Roche-sur-Yon
  - CHRU Lille, Lille
  - CHU Nord Marseille, Marseille
  - CHU Nantes, Nantes
  - CHU Nîmes Caremeau, Nîmes
  - Hôpital Saint-Louis, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Bichat, Paris
  - CH Périgueux, Périgueux
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Sud Réunion, Saint-Pierre
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bertagnolio S, Thwin SS, Silva R, Nagarajan S, Jassat W, Fowler R, Haniffa R, Reveiz L, Ford N, Doherty M, Diaz J. Clinical features of, and risk factors for, severe or fatal COVID-19 among people living with HIV admitted to hospital: analysis of data from the WHO Global Clinical Platform of COVID-19. Lancet HIV. 2022 Jul;9(7):e486-e495. doi: 10.1016/S2352-3018(22)00097-2. Epub 2022 May 10. PMID 35561704
- [Background] DeWolf S, Laracy JC, Perales MA, Kamboj M, van den Brink MRM, Vardhana S. SARS-CoV-2 in immunocompromised individuals. Immunity. 2022 Oct 11;55(10):1779-1798. doi: 10.1016/j.immuni.2022.09.006. Epub 2022 Sep 13. PMID 36182669
- [Background] MacKenna B, Kennedy NA, Mehrkar A, Rowan A, Galloway J, Matthewman J, Mansfield KE, Bechman K, Yates M, Brown J, Schultze A, Norton S, Walker AJ, Morton CE, Harrison D, Bhaskaran K, Rentsch CT, Williamson E, Croker R, Bacon S, Hickman G, Ward T, Davy S, Green A, Fisher L, Hulme W, Bates C, Curtis HJ, Tazare J, Eggo RM, Evans D, Inglesby P, Cockburn J, McDonald HI, Tomlinson LA, Mathur R, Wong AYS, Forbes H, Parry J, Hester F, Harper S, Douglas IJ, Smeeth L, Lees CW, Evans SJW, Goldacre B, Smith CH, Langan SM. Risk of severe COVID-19 outcomes associated with immune-mediated inflammatory diseases and immune-modifying therapies: a nationwide cohort study in the OpenSAFELY platform. Lancet Rheumatol. 2022 Jul;4(7):e490-e506. doi: 10.1016/S2665-9913(22)00098-4. Epub 2022 Jun 9. PMID 35698725
- [Background] Evans RA, Dube S, Lu Y, Yates M, Arnetorp S, Barnes E, Bell S, Carty L, Evans K, Graham S, Justo N, Moss P, Venkatesan S, Yokota R, Ferreira C, McNulty R, Taylor S, Quint JK. Impact of COVID-19 on immunocompromised populations during the Omicron era: insights from the observational population-based INFORM study. Lancet Reg Health Eur. 2023 Oct 13;35:100747. doi: 10.1016/j.lanepe.2023.100747. eCollection 2023 Dec. PMID 38115964